CLINICAL TRIAL: NCT01654666
Title: Protective Effects of Long-term Remote Limb Ischemic Preconditioning For Carotid Artery Stenting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ji Xunming (Other)
Responsible Party: Sponsor-Investigator, Ji Xunming, XuanWu Hospital, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RIPC2012
Record Dates: First submitted 2012-07-23; First posted 2012-08-01 (Estimated); Results first posted 2015-11-11 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-10

CONDITIONS: Carotid Artery Stenosis
Keywords: Remote ischemic preconditioning; Stroke secondary prevention; Carotid artery stenting; Carotid stenosis; Inflammation
MeSH Terms: conditions — Carotid Stenosis; Inflammation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- RIPC group (Experimental): Treatment:Patients in this group received standard medical therapy and remote ischemic preconditioning (RIPC) treatment.
  Device:RIPC consisted of five 5-min cycles of bilateral arm ischemia/reperfusion, which is induced by an automated cuff-inflator placed on bilateral arm and inflated to 200 mmHg for 5-min followed by deflating the cuff for 5-min,each patient in the RIPC group do it twice a day for at least two weeks before carotid artery stenting.
  Procedure: Carotid Artery Stenting
  Interventions: Procedure: Remote ischemic preconditioning; Procedure: Carotid Artery Stenting
- Control group (Active Comparator): Treatment:Patients in this group received standard medical therapy alone. Procedure: Carotid Artery Stenting
  Interventions: Procedure: Carotid Artery Stenting
- Sham RIPC group (Sham Comparator): Treatment:Patients in this group received standard medical therapy and sham remote ischemic preconditioning treatment.
  Device:Sham RIPC consisted of five 5-min cycles of bilateral arm ischemia/reperfusion, which is induced by an automated cuff-inflator placed on bilateral arm and inflated to 60 mmHg for 5-min followed by deflating the cuff for 5-min, each patient in RIPC group do it twice a day for at least two weeks before carotid artery stenting.
  Procedure: Carotid Artery Stenting
  Interventions: Procedure: Sham remote ischemic preconditioning; Procedure: Carotid Artery Stenting

INTERVENTIONS:
Procedure: Remote ischemic preconditioning — Remote ischemic preconditioning consisted of five 5-min cycles of bilateral arm ischemia/reperfusion, which is induced by an automated cuff-inflator placed on bilateral arm and inflated to 200 mmHg for 5-min followed by deflating the cuff for 5-min.
  Other Names: RIPC
  Arms: RIPC group
Procedure: Sham remote ischemic preconditioning — Sham remote ischemic preconditioning consisted of five 5-min cycles of bilateral arm ischemia/reperfusion, which is induced by an automated cuff-inflator placed on bilateral arm and inflated to 60 mmHg for 5-min followed by deflating the cuff for 5-min.
  Other Names: Sham RIPC
  Arms: Sham RIPC group
Procedure: Carotid Artery Stenting — Carotid Artery Stenting is an invasive therapy of carotid artery stenosis.
  Other Names: CAS

SUMMARY:
Remote limb ischemic preconditioning (RIPC) has neuro-protective and anti-inflammatory effects on ischemia- reperfusion injury. As the extent of its effect is unknown, the investigators will use clinical outcome, serum biochemical markers and brain magnetic resonance imaging (MRI) to determine whether RIPC has neuro-protective and anti-inflammatory effects on patients undergoing carotid artery stenting.

DETAILED DESCRIPTION:
BACKGROUND: Brain ischemia and injury contributed to perioperative morbidity and mortality in Carotid Artery Stenting. Remote ischemic preconditioning (RIPC), brief periods of ischemia followed by reperfusion, can provide systemic protection for prolonged ischemia. Our previous study found no significant protection to the patients who received once RIPC before Carotid Artery Stenting. In order to investigate whether long-term RIPC before Carotid Artery Stenting can protect these patients from the perioperative and long-term complications, a prospective randomized controlled trial will be performed in the current study.

DESIGNING: About 189 patients who are eligible for carotid artery stenting will be randomly assigned in 1:1:1 ratio to RIPC group, sham RIPC group and conventional Carotid Artery Stenting group (control). Remote limb ischemic preconditioning (RIPC) is consisted of five 5-min cycles of bilateral arm ischemia/reperfusion, it is induced by an automated cuff-inflator placed on bilateral arm and inflated to 200 mmHg for 5-min followed by deflating the cuff for 5-min, patients in the RIPC group will do it twice a day for at least two weeks before carotid artery stenting. Patients in the sham RIPC group receive sham RIPC treatment, which is consisted of five 5-min cycles of bilateral arm ischemia/reperfusion, induced by an automated cuff-inflator placed on bilateral arm and inflated to 60 mmHg for 5-min followed by deflating the cuff for 5-min, they will do it twice a day for at least two weeks before carotid artery stenting. Patients in the control group receive conventional carotid artery stenting without RIPC or sham RIPC treatment. Cerebral injury is assessed by serum S-100B and Neuron specific enolase (NSE), systematic inflammation is assessed by serum high-sensitivity C-reactive protein (hs-CRP). Post-treatment infarctions, both symptomatic and asymptomatic, are detected by diffusion-weighted imaging (DWI) and clinical outcomes are determined by cerebrovascular events, cardiac events or death.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic or asymptomatic carotid artery stenosis. In symptomatic patients the degree of stenosis should more than 60% (Based on NASCET Criteria), in asymptomatic patients the degree of stenosis should more than 70% (Based on NASCET Criteria);
2. Tolerance to any of the study medications, including clopidogrel, aspirin and statins;
3. Can cooperate with and complete brain MRI examination;
4. Has a negative pregnancy test within 7 days before randomization and no childbearing potential;
5. Vascular ultrasound excluded intravascular thrombosis and unstable plaques in blood vessels of the bilateral upper limbs;
6. No hemorrhagic tendency;
7. Stable vital sign, normal renal and hepatic functions;
8. Informed consent.

Exclusion Criteria:

1. Evolving stroke;
2. Prior major ipsilateral stroke, if likely to confound study endpoints;
3. Severe dementia;
4. Hemorrhagic conversion of an ischemic stroke within the past 60 days;
5. Chronic atrial fibrillation;
6. Myocardial infarction within previous 30 days;
7. Inability to understand and cooperate with study procedures or provide informed consent;
8. Participating in other device or drug trial that has not completed the required protocol follow-up period;
9. Any conditions that hampers proper angiographic assessment or makes percutaneous arterial access unsafe;
10. High risk candidates defined as the Carotid Revascularization Endarterectomy vs. Stenting Trial (CREST);
11. Any vascular, extremity soft tissue or orthopedic injury that may contraindicate bilateral arm ischemic preconditioning (e.g. superficial wounds and fractures of the arm);
12. Blood pressure cannot be controlled lower than 200 mmHg by medications;
13. Peripheral blood vessel disease (especially subclavian arterial and upper limb artery stenosis or occlusion).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2012-07; Primary Completion 2015-01 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji M.D., Ph.D., Principal Investigator — Capital Medical University
Locations (1):
- Baojun Hou, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Liang F, Liu S, Liu G, Liu H, Wang Q, Song B, Yao L. Remote ischaemic preconditioning versus no remote ischaemic preconditioning for vascular and endovascular surgical procedures. Cochrane Database Syst Rev. 2023 Jan 16;1(1):CD008472. doi: 10.1002/14651858.CD008472.pub3. PMID 36645250
- [Derived] Zhao W, Meng R, Ma C, Hou B, Jiao L, Zhu F, Wu W, Shi J, Duan Y, Zhang R, Zhang J, Sun Y, Zhang H, Ling F, Wang Y, Feng W, Ding Y, Ovbiagele B, Ji X. Safety and Efficacy of Remote Ischemic Preconditioning in Patients With Severe Carotid Artery Stenosis Before Carotid Artery Stenting: A Proof-of-Concept, Randomized Controlled Trial. Circulation. 2017 Apr 4;135(14):1325-1335. doi: 10.1161/CIRCULATIONAHA.116.024807. Epub 2017 Feb 7. PMID 28174194

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Symptomatic and asymptomatic subjects with carotid artery stenosis which was more than 70% by angiography , duplex ultrasound, Computed Tomography Angiography or Magnetic Resonance Angiography (NASCET criteria), who could undergo carotid artery stenting and all follow-ups, were recruited starting from August 2012.
Groups:
- RIPC Group: Treatment:Patients in this group received standard medical therapy and remote ischemic preconditioning (RIPC) treatment for at least 2 weeks before carotid artery stenting.
  Remote ischemic preconditioning: Remote ischemic preconditioning consisted of five 5-min cycles of bilateral arm ischemia/reperfusion, which is induced by an automated cuff-inflator placed on bilateral arm and inflated to 200 mmHg for 5-min followed by deflating the cuff for 5-min.
  Carotid Artery Stenting: Carotid Artery Stenting is an invasive therapy of carotid artery stenosis.
- Control Group: Treatment:Patients in this group received standard medical therapy alone for at least 2 weeks before carotid artery stenting.
  Carotid Artery Stenting: Carotid Artery Stenting is an invasive therapy of carotid artery stenosis.
- Sham RIPC Group: Treatment:Patients in this group received standard medical therapy and sham RIPC treatment for at least 2 weeks before carotid artery stenting.
  Sham remote ischemic preconditioning: Sham remote ischemic preconditioning consisted of five 5-min cycles of bilateral arm ischemia/reperfusion, which is induced by an automated cuff-inflator placed on bilateral arm and inflated to 60 mmHg for 5-min followed by deflating the cuff for 5-min.
  Carotid Artery Stenting: Carotid Artery Stenting is an invasive therapy of carotid artery stenosis.
Period: Overall Study
Arm/Group | RIPC Group | Control Group | Sham RIPC Group
Started | 63 | 63 | 63
Primary Analysis | 52 | 56 | 54
Completed | 48 | 50 | 49
Not Completed | 15 | 13 | 14
Not completed — Protocol Violation | 7 | 4 | 8
Not completed — Lost to Follow-up | 4 | 5 | 5
Not completed — Withdrawal by Subject | 4 | 4 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population only included participants who finished carotid artery stenting, post-treatment MRI scans and blood drawn.
Groups:
- Total: Total of all reporting groups
Arm/Group | RIPC Group | Control Group | Sham RIPC Group | Total
Number analyzed (Participants) | 63 | 63 | 63 | 189
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.49 (8.63) | 66.47 (8.54) | 65.71 (8.61) | 66.56 (8.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 19 | 54
  Male | 46 | 45 | 44 | 135
Race/Ethnicity, Customized [Number; unit: participants]
  Han race | 63 | 63 | 63 | 189
Pre-treatment scans [Number; unit: participants]
  New DWI lesions | 2 | 2 | 1 | 5
  No new DWI lesions | 61 | 61 | 62 | 184
Clinical manifestation [Number; unit: participants] — Clinical manifestation of the target carotid artery stenosis.
  participants
    Symptomatic | 41 | 45 | 42 | 128
    Asymptomatic | 22 | 18 | 21 | 61
Contralateral carotid condition [Number; unit: participants]
  Severe stenosis | 5 | 5 | 4 | 14
  Occlusion | 2 | 1 | 2 | 5
  Other | 56 | 57 | 57 | 170

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Cerebrovascular Events, Cardiovascular Events or Death.
Description: Cerebrovascular events included ischemic stroke, transient ischemic attack (TIA), cerebral hemorrhage and hyperperfusion syndrome. Cardiovascular events included angina and myocardial infarction.Death included any reason caused death.
Time Frame: Within six months after carotid artery stenting
Population: The analysis population only included participants who fully completed the study.
Measure: Number; unit: participants
Arm/Group | RIPC Group | Control Group | Sham RIPC Group
Number analyzed (Participants) | 48 | 50 | 49
participants
  Ischemic stroke within 6 months | 0 | 2 | 2
  TIA within 6 months | 1 | 0 | 1
  No cerebrovascular event within 6 months | 47 | 48 | 46
  No Cardiovascular Events | 47 | 48 | 46
  No Deaths | 47 | 48 | 46

2. Primary Outcome: Participants Who Got New Diffusion-weighted Imaging (DWI) Lesions on Post-treatment Magnetic Resonance Imaging (MRI) Scans.
Time Frame: Within 48 hours after carotid artery stenting.
Population: The analysed population only included participants who finished carotid artery stenting, post-treatment MRI scans and blood drawn.
Measure: Number; unit: participants
Arm/Group | RIPC Group | Control Group | Sham RIPC Group
Number analyzed (Participants) | 52 | 56 | 54
participants
  With new lesions on post-treatment scans | 10 | 26 | 23
  Without new lesions on post-treatment scans | 42 | 30 | 31

3. Secondary Outcome: Serum High-sensitive C-reactive Protein (Hs-CRP).
Time Frame: Baseline, on admission, and 1 and 24 hours after carotid artery stenting.
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | RIPC Group | Control Group | Sham RIPC Group
Number analyzed (Participants) | 52 | 56 | 54
mg/L
  Baseline | 1.23 [0.69 to 4.73] | 1.22 [0.76 to 4.67] | 1.37 [0.81 to 3.77]
  On admission | 0.99 [0.59 to 3.51] | 1.09 [0.85 to 2.56] | 1.35 [0.57 to 3.69]
  1 hour after CAS | 1.31 [0.61 to 2.93] | 1.46 [0.78 to 3.60] | 1.55 [1.09 to 4.18]
  24 hours after CAS | 5.09 [2.29 to 11.54] | 7.90 [4.63 to 13.90] | 6.90 [3.75 to 9.72]

4. Secondary Outcome: Number of Patients With Any Side Effects of Remote Ischemic Preconditioning (RIPC) Treatment.
Description: The side effects referred to any side effects of RIPC or sham RIPC treatment, not including the sides effect of medications and CAS.
Time Frame: From baseline to 6 months after treatment.
Measure: Number; unit: participants
Arm/Group | RIPC Group | Control Group | Sham RIPC Group
Number analyzed (Participants) | 48 | 50 | 49
participants | 0 | 0 | 0

5. Secondary Outcome: Serum Neuron Specific Enolase (NSE) Levels.
Time Frame: Baseline, on admission, and 1 and 24 hours after carotid artery stenting.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | RIPC Group | Control Group | Sham RIPC Group
Number analyzed (Participants) | 52 | 56 | 54
ng/L
  Baseline | 12.83 (3.07) | 12.51 (2.92) | 12.12 (2.76)
  On admission | 12.63 (3.77) | 12.85 (3.59) | 12.56 (2.71)
  1 hour after CAS | 13.00 (2.85) | 13.18 (3.98) | 13.01 (4.32)
  24 hours after CAS | 12.65 (2.78) | 12.97 (4.28) | 12.77 (3.05)

6. Secondary Outcome: Serum S-100B Levels.
Time Frame: Baseline, on admission, and 1 and 24 hours after carotid artery stenting.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | RIPC Group | Control Group | Sham RIPC Group
Number analyzed (Participants) | 52 | 56 | 54
pg/mL
  Baseline | 49.64 (15.74) | 50.14 (17.04) | 50.42 (13.62)
  On admission | 49.70 (16.25) | 50.75 (16.79) | 51.24 (13.30)
  1 hour after CAS | 50.99 (20.21) | 51.19 (22.40) | 51.79 (19.42)
  24 hours after CAS | 51.40 (16.16) | 52.94 (24.34) | 52.02 (19.71)

ADVERSE EVENTS:
Time Frame: Through 6 months post carotid artery stenting.
Arm/Group | RIPC Group | Control Group | Sham RIPC Group
Serious Adverse Events (participants affected / at risk) | 1/52 | 3/56 | 3/54
Other Adverse Events (participants affected / at risk) | 10/52 | 26/56 | 23/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RIPC Group (N=52) | Control Group (N=56) | Sham RIPC Group (N=54)
Hyperperfusion Syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — The hyperperfusion syndrome is characterized by headache, focal motor seizures and intracerebral hemorrhage, it can be evidenced by head Computed Tomography, Magnetic Resonance Imaging, Electroencephalogram.
Symptomatic Ischemic Stroke (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) — Symptomatic ischemic stroke is defined as an acute neurological event lasting over 24 hours with focal signs and symptoms
Transient Ischemic Attack (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) — Transient ischemic attack (TIA) is a brief episode (<24 hours) of neurologic dysfunction resulting from focal temporary cerebral ischemia not associated with cerebral infarction.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RIPC Group (N=52) | Control Group (N=56) | Sham RIPC Group (N=54)
At least one new lesion (Nervous system disorders) | 10 (10) | 26 (26) | 23 (23) — Number of participant with new DWI lesions on post-treatment MRI scans

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No